CLINICAL TRIAL: NCT04252196
Title: Arm Motor Rehabilitation, Entertainment and Cognition System for the Elderly (Usability Study)
Brief Title: Arm Motor Rehabilitation, Entertainment and Cognition System for the Elderly.BAC.U
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bright Cloud International Corp (Industry)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Dr. Nam H. Kim, Director of Engineering, Bright Cloud International Corp
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BCI-10-001.BAC.U; 5R44AG044639-05 (NIH)
Record Dates: First submitted 2020-01-22; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Device usability single group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Device Usability Study (Experimental): Usability evaluators of medical device (Healthy volunteers).
  Interventions: Device: usability evaluation of medical device

INTERVENTIONS:
Device: usability evaluation of medical device — participants interact with medical device and rate it for usability

SUMMARY:
This usability study is to test the basic functionality of the BrightArm Compact (BAC) system. The BAC is a motorized rehabilitation platform to offer gravity bearing for weak upper extremity. It has a medical grade PC which hosts numerous interactive, adaptable computer games, played using BrightBrainer Grasp (BBG) controllers. The device is passive, in that no actuators apply forces on the patient. Further, the patient is free to lift that arm, nothing restricts the arms movement away from the BAC table.

DETAILED DESCRIPTION:
Healthy, age matched participants are invited to test the BAC at Bright Cloud Int Corporate Labs (675 US Hwy 1 south, B203, North Brunswick, NJ 08902, USA).

At the beginning of the usability training, participants will be required to sign a consent form, and BCI research staff will go over the details of the study and check inclusion criteria (generally healthy individual, age 50 ~ 85, English speaker, cognitively normal).

Subjects participate in 4 study sessions over approximately 1 month, each session lasting about an hour. The BAC table will have a different configuration each session. In the first session the table will have 0 tilt (flat). In session 2 it will be tilted 10 degrees downwards, in session 3 the table will be tilted up 10 degrees and in Session 4 the BAC table will be tilted up 20 degrees.

The difficulty of the games will also vary from session to session, progressing from the lowest difficulty in Session 1 to the highest difficulty in Session 4. Thus a given game will not be exactly the same, when played in a subsequent session, so to allow varying interaction scenarios.

At the end of each session, participants will be asked to fill up a custom feedback form. The custom form has questions on the system, the rehabilitation table, the controller, the therapeutic games they tested, and their overall impression of the experimental device. Each question on the custom form is answered on a 5-point Liker Scale.

At the end of the last session they will fill a standardized USE form, with questions rated on a 7-point Likert scale.

Feedback from participant will be used to improve the device as well as the therapeutic games.

ELIGIBILITY:
Inclusion Criteria:

* generally healthy
* age 50~80;
* good or corrected vision;
* good or corrected hearing

Exclusion Criteria:

* motor or cognitively impaired;
* outside 50~80 age bracket;
* inability to speak English;
* history of violence or drug abuse.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2019-01-28 (Actual); Study Completion 2019-01-28 (Actual)

PRIMARY OUTCOMES:
Subjective evaluation of medical device (custom questionnaire) | 4 weeks
  Custom questionnaire rating on a 5 point Likert scale. 1 (min), 5 (max), larger number means better outcomes
USE Questionnaire | 1 weeks
  Participants fill the standardized USE questionnaire rating the BrightArm Compact system on a 7-point Likert Scale. 1 (min), 7 (max), larger number means better outcomes.

SECONDARY OUTCOMES:
Game errors | 4 weeks
  Participants play a number of custom, adaptable therapeutic games, and their errors are stored. Min number is 0, which is also the best outcome.
Game difficulty | 4 weeks
  Participants play a number of custom, adaptable therapeutic games, and their game difficulty level is stored each time. Min is 1, larger number is better
Game scores | 4 weeks
  Participants play a number of custom, adaptable therapeutic games, and their game scores are stored each time. Min score is 0, larger score is better.
Level of comfort | 4 weeks
  Participants play a number of custom, adaptable therapeutic games, at varying device configuration and report on perceived level of comfort (free form).
Device ruggedness | 4 weeks
  Participants play a number of custom, adaptable therapeutic games, at varying device configuration and report on frequency of technical issues (free form).

CONTACTS AND LOCATIONS:
Locations (1):
- Commercialization Center for Innovative Technologies, Suite B203, North Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BCI's corporate site showing BrightArm device development — http://www.brightcloudint.com

DOCUMENTS (2):
  • Informed Consent Form (2018-09-05): https://cdn.clinicaltrials.gov/large-docs/96/NCT04252196/ICF_000.pdf
  • Study Protocol (2018-08-24): https://cdn.clinicaltrials.gov/large-docs/96/NCT04252196/Prot_001.pdf